CLINICAL TRIAL: NCT06455826
Title: A Phase 1 Open-Label, Multiple Ascending Dose Study to Evaluate the Safety and Tolerability of Intravitreally Administered VP-001 in Participants With Confirmed PRPF31 Mutation-Associated Retinal Dystrophy
Brief Title: MAD of IVT VP-001 in PRPF31 Mutation-Associated Retinal Dystrophy Subjects (Wallaby)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: PYC Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: VP001-CL102
Record Dates: First submitted 2024-06-03; First posted 2024-06-12 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Retinitis Pigmentosa 11; Retinal Degeneration; Eye Diseases; Retinal Disease; Retinal Dystrophies
MeSH Terms: conditions — Retinitis Pigmentosa 11; Retinal Degeneration; Eye Diseases; Retinal Diseases; Retinal Dystrophies

STUDY DESIGN:
Intervention Model Description: Participants will be assigned sequentially to the VP-001 escalation dose (30 μg and 75 μg) groups. Participants will receive three repeat IVT injections of VP-001, 8 weeks apart, in the study eye.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Multi-ascending dose escalation study of VP-001 (Experimental)
  Interventions: Drug: VP-001

INTERVENTIONS:
Drug: VP-001 — A Phase 1 Open-Label, Multiple Ascending Dose Study of VP-001 in Participants with Confirmed PRPF31 Mutation- Associated Retinal Dystrophy

SUMMARY:
A Phase 1 Open-Label, Multiple Ascending Dose Study to Evaluate the Safety and Tolerability of Intravitreally Administered VP-001 in Participants with Confirmed PRPF31 Mutation-Associated Retinal Dystrophy

ELIGIBILITY:
Inclusion Criteria:

1. Male or female sex; ≥12 years of age at Baseline (Visit 2).
2. Have a molecular (genetic) diagnosis of PRPF31 mutation.
3. Have a clinical diagnosis of PRPF31 mutation-associated retinal dystrophy, that is, RP11. The following conditions are allowed for inclusion if due to RP11, if in the opinion of the investigator they will not interfere with study evaluations or have resolved: macular edema (intraretinal, sub-retinal or other fluid) requiring regular treatment at a frequency of less than every 6 weeks; macular edema must be stable for at least 3 months prior to Screening (Visit 1). The investigator must consult with the study Medical Monitor.
4. If ≥18 years of age, understand the language of the informed consent and are willing and able to provide written informed consent prior to any study procedures. If a minor (12 to <18 years of age), a parent or legal guardian willing and able to provide written permission for the minor's participation prior to performing any study related procedures and pediatric participant able to provide age appropriate assent for study participation.
5. If ≥18 years of age, are willing to comply with the instructions and attend all scheduled study visits. If a minor (12 to <18 years of age), able to complete all study assessments, comply with the protocol, and has a parent or caregiver willing and able to follow study instructions and attend study visits with the participant as required, in the opinion of the Investigator.
6. Meets ≥1 of the following for visual function in the study eye:

   1. V4e visual field >1000 deg2, per kinetic perimetry
   2. <Mean microperimetry threshold: >5 decibel (dB) to <15dB
   3. Visual acuity: 20/40 to 20/200 inclusive (>35 and <70 letters by Early-Treatment Diabetic Retinopathy Study [ETDRS])
   4. Ellipsoid zone (EZ) length >1000 microns, of which 500 microns is contiguous, by SD-OCT
   5. FST baseline no worse than -20 dB
7. Participants of childbearing potential and male participants must not be pregnant or lactating and must be sexually inactive by abstinence, which is consistent with the preferred and usual lifestyle of the participant or agree to use adequate birth control throughout study duration. Adequate birth control is defined as hormonal - oral, implantable, injectable, or transdermal contraceptives; mechanical - spermicide in conjunction with a barrier such as a condom or diaphragm; intrauterine device (IUD); or surgical sterilization of partner. For nonsexually active participants, abstinence may be regarded as an adequate method of birth control. Participants of childbearing potential include all participants who have experienced menarche and have not undergone successful surgical sterilization (bilateral tubal ligation, hysterectomy, or bilateral oophorectomy) or are not postmenopausal (12 months after last menses).

Exclusion Criteria:

1. Have any uncontrolled systemic disease that, in the opinion of the Investigator, would preclude participation in the study that include but are not limited to infection, uncontrolled elevated blood pressure, cardiovascular disease, or glycemic control issues, or any other medical condition that may put the participant at risk due to study procedures.
2. Mutations in genes that cause autosomal dominant RP, Xlinked RP, or presence of biallelic mutations in autosomal recessive RP/retinal dystrophy genes other than PRPF31 mutations.
3. Have used anti-vascular endothelial growth factor (VEGF) agents within 2 months or corticosteroid injections within the last 3 months.
4. Have had Ozurdex

   * implants placed within 3 months or Retisert
   * or Iluvien
   * implants placed within 3 years prior to Baseline (Visit 2).
5. Within 3 months prior to Baseline (Visit 2), have undergone any vitreoretinal surgery (scleral buckle, pars plana vitrectomy, retrieval of a dropped nucleus or intraocular lens, radial optic neurotomy, sheathotomy, cyclodestructive procedures or multiple filtration surgeries [2 or more]) or any other ocular surgery.
6. Have ocular media opacity or poor pupillary dilation prohibiting quality ophthalmic evaluation or photography, as assessed by the investigator.
7. Have used any investigational drug or device within 90 days or 5 estimated half-lives of Baseline (Visit 2), whichever is longer, or plan to participate in another study of drug or device during the study period. Participation in observational trials is allowable based on investigator discretion and consultation with the Medical Monitor. It is assumed that the observational trial evaluations would not interfere with participation in this study.
8. Have received any prior cell, ribonucleic acid (RNA) (including VP-001), or gene therapy for a retinal condition.
9. Have a recent history (<6 months) or current excessive recreational drug or alcohol use, in the opinion of the investigator.
10. Any retinal pathology other than RP11 that in the investigator's opinion could affect study results.
11. Participants should not have any conditions, in the investigator's opinion, that may put the participant at increased risk, confound study data, or interfere significantly with the participant's study participation.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-06-13 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
The incidence, severity, and relatedness of treatment-emergent ocular adverse events and treatment-emergent serious adverse events | over a 4-week post-dose period
The incidence, severity, and relatedness of treatment-emergent ocular adverse events | over a 52-week period

SECONDARY OUTCOMES:
Adverse Events and Treatment Emergent serious adverse events (TESAEs) in the fellow eye eye | over a 4-week post-dose time period
Adverse Events and Treatment Emergent serious adverse events (TESAEs) in the fellow eye eye | over a 52-week period
Incidence, severity, and relatedness of non-ocular Treatment Emergent adverse events (TEAEs) | over a 4-week post-dose time period
Incidence, severity, and relatedness of non-ocular Treatment Emergent adverse events (TEAEs) | over a 52-week period
BCVA letter score using ETDRS charts | over a 52-week period
Change in lowest passing light level using Ora- VNC™ mobility test | over a 52-week period
Low luminance visual acuity (LLVA) letter score | over a 52-week period
Visual field sensitivity as measured by static perimetry with topographic analysis (Hill of Vision) | over a 52-week period
Mean retinal sensitivity as measured by fundusguided microperimetry | over a 52-week period
Visual fields as measured by kinetic perimetry utilizing I4e, II4e and V4e stimuli | over a 52-week period
Rod-and cone-mediated retinal function as measured by white, red and blue FST | over a 52-week period
Retinal thickness on SD-OCT, including retinal thickness in each ETDRS subfield and EZ area and volume | over a 52-week period
Retinal function using full-field electroretinography (ERG) | over a 52-week period
Area of hypo-autofluorescence captured by FAF | over a 52-week period
Abnormalities captured by wide-field fundus photography | over a 52-week period

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - University of Florida Health, Jacksonville, Florida
  - University of Michigan Kellogg Eye Center, Ann Arbor, Michigan
  - Oregon Health and Science University - Casey Eye Institute, Portland, Oregon
  - Retina Foundation of the Southwest, Dallas, Texas
  - Baylor College of Medicine- Alkek Eye Center, Houston, Texas